CLINICAL TRIAL: NCT04903392
Title: Investigation of the Effects of Gait Training on Balance, Plantar Pressure Distribution and Respiratory Parameters in Chronic Stroke Patients
Brief Title: Effects of Backward Gait Training in Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Burçin Akçay, Assistant Professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAkcay
Record Dates: First submitted 2021-05-18; First posted 2021-05-26 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Chronic Stroke Patients
Keywords: Chronic Stroke Patients; Balance; Plantar Pressure Distribution; Respiratory Parameters; Backward Gait Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Backward Walking Group (Experimental): Conventional therapy + Backward Walking Training
  Interventions: Other: Backward Walking Training
- Forward Walking Group (Other): Conventional therapy + Forward Walking Training
  Interventions: Other: Forward Walking Training

INTERVENTIONS:
Other: Backward Walking Training — The training speed will start at the basic walking speed and will increase by 5% of the starting speed each week. The training, which will take 30 minutes, will be as follows: 5 minutes forward walking (warm-up phase), 20 minutes backward walking (intervention phase) and 5 minutes forward (cooling phase).
  -three times a week for six weeks
  Arms: Backward Walking Group
Other: Forward Walking Training — The training speed will start at the basic walking speed and will increase by 5% of the starting speed each week. It will be in the form of walking forward for 30 minutes.
  -three times a week for six weeks
  Arms: Forward Walking Group

SUMMARY:
Loss of motor control after stroke, muscle weakness, abnormal movement patterns, spasticity, range of motion limitations and sensory dysfunction, resulting in a decrease in the load transferred to the affected limb, changes in gait pattern and balance skills. Post-stroke muscle weakness has been shown to occur not only in the lower and upper extremity muscles but also in the respiratory muscles. It was found that the plantar pressure distribution in the affected side feet was decreased in individuals with stroke and this situation negatively affected the walking function. A systematic review of treadmill training revealed that treadmill training significantly increased walking speed and walking distance. Learning to walk backwards is also recommended to improve the movement components required for walking forward. As a result of the investigations, although there are studies about the effects of back-walking training on walking and balance function in chronic stroke patients, there is no study investigating the effects on plantar pressure distribution and respiratory parameters. Therefore, this study, which planned to investigate the effects of treadmill retching training on balance, plantar pressure distribution and respiratory parameters in chronic stroke patients, will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* More than 6 months have passed since the onset of stroke
* First time stroke diagnosis
* Being between the ages of 40-65
* Spasticity severity in lower extremity less than 3 according to Modified Ashworth Scale,
* Being medically stable
* Ability to walk 10 meters and above without assistance

Exclusion Criteria:

* Presence of other neurological or orthopedic diseases that affect standing and walking involving the lower limbs
* Uncontrollable Hypertension
* Having been diagnosed with any pulmonary disease
* Severe cardiac conditions
* Uncontrollable DM
* Lack of cooperation

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Plantar pressure assessment | 6 weeks
  Plantar pressure distribution will be evaluated.
Balance assessment | 6 weeks
  Static and dynamic balance will be evaluated with The Korebalance Premiere device.
Pulmonary function (Forced vital capacity (FVC)) | 6 weeks
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced vital capacity (FVC) will be evaluated.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | 6 weeks
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced expiratory volume in the first second (FEV1) will be evaluated.
Pulmonary function (FEV1 / FVC) | 6 weeks
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, FEV1 / FVC will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | 6 weeks
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Pulmonary function (Peak flow rate (PEF)) | 6 weeks
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, peak flow rate (PEF) will be evaluated.
Respiratory Muscle Strength | 6 weeks
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be measured using portable, electronic, oral pressure measuring device

CONTACTS AND LOCATIONS:
Locations (1):
- Burçin Akçay, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim KH, Lee KB, Bae YH, Fong SSM, Lee SM. Effects of progressive backward body weight suppoted treadmill training on gait ability in chronic stroke patients: A randomized controlled trial. Technol Health Care. 2017 Oct 23;25(5):867-876. doi: 10.3233/THC-160720. PMID 28759977
- [Background] Munari D, Serina A, Disaro J, Modenese A, Filippetti M, Gandolfi M, Smania N, Picelli A. Combined effects of backward treadmill training and botulinum toxin type A therapy on gait and balance in patients with chronic stroke: A pilot, single-blind, randomized controlled trial. NeuroRehabilitation. 2020;46(4):519-528. doi: 10.3233/NRE-203067. PMID 32508341
- [Background] Nadeau S, Amblard B, Mesure S, Bourbonnais D. Head and trunk stabilization strategies during forward and backward walking in healthy adults. Gait Posture. 2003 Dec;18(3):134-42. doi: 10.1016/s0966-6362(02)00070-x. PMID 14667946
- [Background] Weng CS, Wang J, Pan XY, Yu ZZ, Wang G, Gao LP, Huo CN. [Effectiveness of backward walking treadmill training in lower extremity function after stroke]. Zhonghua Yi Xue Za Zhi. 2006 Oct 10;86(37):2635-8. Chinese. PMID 17198591
- [Background] Yang YR, Yen JG, Wang RY, Yen LL, Lieu FK. Gait outcomes after additional backward walking training in patients with stroke: a randomized controlled trial. Clin Rehabil. 2005 May;19(3):264-73. doi: 10.1191/0269215505cr860oa. PMID 15859527